CLINICAL TRIAL: NCT03105232
Title: Opioid-Redox Study
Acronym: ORS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pavol Jozef Safarik University (Other)
Collaborators: F.D. Roosevelt Teaching Hospital with Policlinic Banska Bystrica (Other)
Responsible Party: Principal Investigator, Kočan Ladislav, MD Ladislav Kočan PhD, Pavol Jozef Safarik University
Other Study IDs: N28/11/16
Record Dates: First submitted 2017-04-02; First posted 2017-04-07 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Opioid Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Group A: Morphin, Hydromorfon, Oxycodon
- Group B: Buprenorfin
- Group C: Fentanyl
- Group D: Opioid rotation

SUMMARY:
Side effects of opioids can from practical view be divided into short-term and long-term. Nervous system disorders are manifested by psychological status changes of the patient and may cause confusion, mental and somatic dependency, dizziness and so on. Influencing the vegetative and cardiovascular system hypotension can occur what is manifestation of vasodilation and decreased myocardial inotropic activity. Another clinical sign is bradycardia and is characterized by general weakness, sweating, collapse can develop. Effects of opioids may cause respiratory depression, bronchospasm and bronchoconstriction. Side effects on the gastrointestinal tract are nausea, vomiting, constipation and less frequently dry mouth. The constipation does not develop tolerance and has to be avoided (dietary modification, laxatives prevention) respectively during long-term opioid treatment obstipation should be affected by blocking peripheral opioid receptors in the gastrointestinal tract by application of an opioid antagonist methylnaltrexone, which does not cross the blood brain barrier, or using naloxone, which is metabolized by "first-pass" metabolism in the liver for example combined preparation containing oxycodone and naloxone (Kulichová, 2012). Known side effects on parenchymatous organ especially on liver is restricted biliary excretion caused by spasm of the biliary tract. Skin manifestations caused by the effects of opioids are urticaria, dermatitis, and pruritus. Renal and urinary disorders may develop as urinary retention and ureteral spasm. Rarely can occur disorders of the immune system, which through the development of hypersensitivity may lead to the development of anaphylactic shock (Kulichová, 2012). Opioids have a negative effect and the endocrine system. Various studies have demonstrated the influence of opioids on regulatory mechanisms. Fundamental changes occur in hypothalamic-pituitary complex, which directs the activities of all the endocrine system. Secretion of hormones of the pituitary gland regulates the nervous system through the hypothalamus, which is the coordination center of autonomic function. The pituitary gland has coordinating function in relation to other endocrine glands, and by production of their hormones affects the peripheral endocrine organs and the targeting tissues (Kulichová, 2012), (Colameco, 2009).

Opioids decrease the secretion of gonadotropin-stimulating hormone, resulting in reduced levels of luteinizing hormone. The result of these changes is reduced secretion of testosterone and estradiol what results in symptoms of hypogonadism. Chronic administration of exogenous opioids decreases the levels of adrenocorticotropic hormone and cortisol, as well as their circadian rhythms. The result is a reduction in the response to stress. Effect on prolactin is not entirely clear. Opioids can stimulate the hypothalamus through the thyroid stimulating hormone, which may cause prolonged and increased response to opioids in patients with hypothyroidism. Chronic use of opioids is associated with weight gain, hyperglycemia and diabetes can worsen (Kulichová, 2012). It may be related to central effects through the sympathetic nervous system and impaired insulin secretion. New laboratory measurements show the development of oxidative stress in patients receiving morphine and related drugs (Merdin, 2016).

The consequences of these biochemical changes further negatively affect the clinical outcome of the patients. They may become predisposed to excessive progression of previously latent diseases whose manifestations in patients previously were not apparent and there is emergence of new diseases. The present data are essential to create a clinical prospective observational studies to clarify this issue and its conclusions would be essential for new therapeutic options for adjuvant therapy in patients suffering from chronic pain.

DETAILED DESCRIPTION:
The process of the study, the choice of the patients, the collection and the processing of data A. Potential participants of study will be familiarized with the course of research in every detail before entering the study and after signing of an informed consent they will be examined by algesiologist. The patients will receive ID number generated by computer because of preserving of anonymity for the purpose of statistical processing of the data. Monitored clinical parameters: The current consumption of analgesics, examination of the type of pain (nociceptive vs. neuropathic - completed questionnaire for PainDetect, DN4 and LANSS Pain scales), demographic information (weight, height, age). Examination of biochemical parameters (ALT, AST, GMT, bilirubin, urea, creatinine, creatinine clearance, antioxidant enzymes and their substrates (glutathione peroxidase, glutathione reductase, catalase, superoxide dismutase, glutathione). These data will be entered into an online database. The statistical analysis of the activities of the enzymes will determine the confidence interval (CI) of 95%. Patients whose entrance numbers will be in this range will keep on in the study, remaining patients will be excluded. The patients who will keep on in study will be divided into four groups.

Group A: patients with chronic pain taking morphine, hydromorphone, oxycodone Group B: patients with chronic pain taking transdermal patch (Buprenorphine) Group C: patients with chronic pain taking transdermal patch (Fentanyl) Group D: opioid rotation B. The first inspection will be carried out 6 months after the beginning of taking of opioids for severe pain. During the first inspection, clinical and biochemical parameters will be examined same as during the input examination of the patient. The patient will fill out a questionnaire PainDetect, DN4 and LANSS Pain scales. C. The second inspection will be carried out 12 months after the beginning of taking of opioids for severe pain. During the second inspection, clinical and biochemical parameters will be examined same as during the previous two patient examinations. The patient will fill out a questionnaire PainDetect, DN4 and LANSS Pain scales.

ELIGIBILITY:
Inclusion Criteria:

* opiod therapy

Exclusion Criteria:

* active chemotherapy or radiotherapy

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with chronic pain who start opioid longterm therapy
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-20 (Estimated); Primary Completion 2021-11-21 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Antioxidant enzymes | 2 years
  SOD, CAT, GPX, Glutation reduktase, glutathion

SECONDARY OUTCOMES:
Numerical pain scale | 2 years
  clinical outcome
Pain detetct score | 2 years
  clinical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Janka Vašková, MD PhD, Principal Investigator — Pavol Jozef Šafárik University in Kosice; Jana Šimonová, MD PhD, Study Chair — Louis Pasteur University Hospital in Košice; Daniela Ogurčáková, MD PhD, Study Chair — Pavol Jozef Šafárik University in Kosice; Peter Čandík, MD PhD, Study Chair — East Slovak Institute of Cardiovascular Disease in Kosice
Locations (1):
- 1st clinic of anesthesiology and intesive care, University hospital of Louis Pasteur, Košice, Slovakia

IPD SHARING:
Plan to Share IPD: No